CLINICAL TRIAL: NCT01121770
Title: Pharmacokinetic Study of Fondaparinux in Inpatients With Renal Dysfunction
Brief Title: "Pharmacokinetic Study of Fondaparinux in Inpatients With Renal Dysfunction"
Acronym: FONDA PK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00021052; 112972
Record Dates: First submitted 2010-05-06; First posted 2010-05-12 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — Fondaparinux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arixtra (Experimental)
  Interventions: Drug: fondaparinux sodium injection

INTERVENTIONS:
Drug: fondaparinux sodium injection — 1.5mg subcutaneously every day

SUMMARY:
The purpose of this study is to determine a preventative dose of study drug, Arixtra® for patients with kidney disease. We will measure the blood levels of Arixtra® in patients with kidney disease and develop guidelines for dosing.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients who are 18 years or older
* estimated creatinine clearances between 20-50 ml/min
* current hospitalization for a cancer-related abdominal, breast surgery or elective orthopedic surgery
* able to give informed consent
* need for prophylactic anticoagulant therapy for increased risk of a thrombotic episode

Exclusion Criteria: Use of the following

* clopidogrel, aspirin, or NSAID usage,(usage is prohibited while patients are participating in the study)
* body weight < 50 kg
* anticoagulation therapy for thrombosis or other indication
* pregnant or breast-feeding
* hypersensitivity to Arixtra®
* thrombocytopenia associated with a positive in vitro test for anti-platelet antibody in the presence of Arixtra®
* bacterial endocarditis
* brain malignancy
* increased risk of bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-05; Primary Completion 2012-10 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Blood samples to measure specific Arixtra® concentration | • Three blood samples for PK analyses will be obtained within the 24 hour period immediately following either the third or fourth consecutive dose of Arixtra
  peak level will be collected 2-3 hours after the dose interval level will be collected between peak and midpoint midpoint level will be collected 12 hours after the dose interval level will be collected midpoint and trough trough level will be collected just prior to the next scheduled dose

SECONDARY OUTCOMES:
Frequency of bleeding events and new thrombotic events | Daily assessments will be made for bleeding and thrombosis
  events will be used to compare to rates in patients without renal dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L Ortel, M.D, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- See also: The Duke Hemostasis & Thrombosis Center provides a multidisciplinary approach to the diagnosis and management of a wide variety of hemostatic disorders and is a leader in basic research effort. Click here for more information about this study. — http://htc.medicine.duke.edu/